CLINICAL TRIAL: NCT01984281
Title: Effects of a Pedometer-based Unsupervised Exercise Program Upon Lifestyle Physical Activity of Asthmatic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Principal Investigator, Cristina Martins Coelho, MSc, Federal University of Juiz de Fora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 13804413.3.1001.5133
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: Physical Activity; Pedometers; Quality of Life
MeSH Terms: conditions — Asthma; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pedometer-based prescription (Experimental): After baseline assessments, the control group will receive a educational session, regarding important aspects of asthma (symptoms, treatment, exacerbations, triggers, etc) plus a unsupervised exercise prescription (walking, 5 times per week, for at least 30 minutes) and a pedometer-based physical activity prescription, consisting of targets to be achieved (in terms of steps per day).
  Interventions: Behavioral: Pedometer-based physical activity prescription
- Control (No Intervention): After baseline assessments, the control group will receive a educational session, regarding important aspects of asthma (symptoms, treatment, exacerbations, triggers, etc) plus a unsupervised exercise prescription (walking, 5 times per week, for at least 30 minutes).

INTERVENTIONS:
Behavioral: Pedometer-based physical activity prescription — After baseline assessments, both groups will receive a educational session, regarding important aspects of asthma plus a unsupervised exercise prescription (walking, 5 times per week, for at least 30 minutes). Only the experimental group will receive a pedometer-based physical activity prescription, consisting of targets (steps per day) to be achieved. The initial target will be determined based on the average of steps per day assessed during the baseline assessments plus 1000 steps. The targets will be biweekly. Both groups will be contact once a week (by phone) and will be asked to return for asthma control assessments once a month.
  Arms: Pedometer-based prescription

SUMMARY:
The purpose of this study is to determine whether a pedometer-based unsupervised exercise program is more effective than a general exercise recommendation to increase lifestyle physical activity in adult patients with asthma.

DETAILED DESCRIPTION:
The patients will be randomized in two groups: the intervention group will receive a standardized advice to physical activity practice plus pedometers and step goals to achieve over the next twelve weeks and the control group will receive the same standardized advice to physical activity practice and usual care.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis for at least 6 months (according to Global Initiative for Asthma criteria)
* Regular drug therapy (inhaled corticosteroids or inhaled corticosteroids plus long-acting beta-agonists)
* Clinical stability during the run-in period (3 weeks)

Exclusion Criteria:

* Physical activity practice over once a week
* Disabling musculoskeletal disease
* Cardiopathy
* Other lung disease
* More than 10 pack-years of smoking
* Pregnancy
* Refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Lifestyle physical activity | 12 weeks
  The lifestyle physical activity will be estimated as the mean number of steps taken in six days using a pedometer (SW200, YAMAX,Tokyo, Japan)

SECONDARY OUTCOMES:
Exercise capacity | 12 weeks
  Exercise capacity will be assessed through the six-minute walking teste.
Asthma Health related quality of life | 12 weeks
  Asthma Health related quality of life will be assessed through the Asthma Quality of Life Questionnaire.
Asthma Control | 12 weeks
  Asthma Control will be assessed through the Asthma Control Questionnaire
Depression and anxiety | 12 weeks
  Depression and anxiety will be assessed through the Hospital Anxiety and Depression Scale
Asthma exacerbations | 12 weeks
  Asthma exacerbations will be assessed through exacerbation diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno V Pinheiro, DSc, Study Director — Federal University of Juiz de Fora; Cristina M Coelho, MSc, Principal Investigator — Federal University of Juiz de Fora
Locations (1):
- University Hospital of the Federal University of Juiz de Fora, Juiz de Fora, Minas Gerais, Brazil